CLINICAL TRIAL: NCT04488068
Title: Feasibility Testing of Transpelvic Magnetic Stimulation as a Novel Intervention toImprove Urogenital Function in Prostate Cancer Survivors
Brief Title: Transpelvic Magnetic Stimulation to Improve Urogenital Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F3455-P
Record Dates: First submitted 2020-06-29; First posted 2020-07-27 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer; Erectile Dysfunction
Keywords: urinary incontinence; hemodynamics
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Intervention to prevent prostate cancer surgery related urological issues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnetic Stimulation (Experimental): Patients will be subjected to TPMS.
  Interventions: Procedure: Sham Magnetic stimulation
- Sham TPMS (No Intervention): Patients will be subjected to sham TPMS

INTERVENTIONS:
Procedure: Sham Magnetic stimulation — Sham Magnetic stimulation for comparison.
  Arms: Magnetic Stimulation

SUMMARY:
After recruitment, 20 male patients will be assigned 1:1 to either age-matched control (G1: sham) or age-matched intervention (G2: pelvic magnetic stimulation; TPMS) groups using computer-generated process, and baseline parameters will be established. All patients will be instructed by the investigators to perform standard of care pelvic floor exercise for the duration of the study. In addition, G2 patients will receive TPMS, while G1 patients will undergo sham treatment.

DETAILED DESCRIPTION:
The investigators will use a custom TPMS device that targets pelvic muscles. The investigators will apply low amplitude (5%) TPMS to improve blood flow, then high amplitude (30-50%) to strengthen pelvic muscles. The treatment regimen will involve two 20-minute sessions/visit and 2 -visits per week for 12-weeks (final monitoring at 24 weeks). TPMS will be administered by a trained clinical coordinator under the supervision of a urologist. Symptom scores and hemodynamic changes will be evaluated monthly. MRI for assessing muscle thickness will be performed in the beginning (before TPMS) and at the end (after TPMS) of the study. The investigators will assess functional improvements using symptom scores. Morphological changes will be determined by MRI.

The secondary outcome measures: Change in number of pads used as a measure of Improvements in continence function, Improvements in penile blood flow change, Improvements in pelvic muscle thickness change, Change in Pad weight as a measure of Improvements in continence function; were changed/replaced by secondary outcome measures that clearly align with the proposed aims of the study as follows: 1) To show the feasibility of recruitment of prostate cancer survivors, acceptability of Transpelvic magnetic Stimulation (TPMS) intervention, and retention of this Veteran population, we will demonstrate recruitment in VA SAN DIEGO HEALTH CARE SYSTEM (VASDHS) urology clinics and retention of these patients for the study duration. 2) To test the feasibility of administering symptom scores in this population to detect severity and early recovery of functional impairment. 3) To test the feasibility of diagnostic imaging to establish: penile/ pelvic floor muscle (PFM) blood flow, PFM anatomical and morphological changes before surgery, immediately after surgery, and after TPMS interventions.

The third aim of the study was not feasible as the study was performed during the pandemic. Therefore, the outcome measures: Improvements in penile blood flow change and Improvements in pelvic muscle thickness change were removed. The secondary outcome measures were to test the feasibility of administering symptom scores in this population of prostate cancer survivors (not efficacy). Therefore, the outcome measures: Change in number of pads used as a measure of Improvements in continence function and Change in Pad weight as a measure of Improvements in continence function were removed. The secondary outcome measures were changed to the current outcome measures: Number of Patients that completed The International Consultation on Incontinence Questionnaire (ICIQ) scores (as a measure of urinary incontinence; UI ) and Number of Patients that completed The International Index of Erectile Function (IIEF; as a measure of erectile dysfunction; ED) scores as these measures directly align with our study aims. Final monitoring at 24 weeks also was not feasible, so the outcome measure time frame was 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* men over 50 years old who are enrolled for prostate surgery,
* have serum testosterone within normal limits, and
* are without prior bilateral orchiectomy, chemotherapy, external radiotherapy, brachytherapy, surgical, or other ablative therapy for prostate cancer.

Exclusion Criteria:

* patients with ED caused by psychological, neurogenic (after non-nerve sparing prostate surgery), or hormonal disorders,
* patients with genital abnormalities precluding intercourse, prior penile implantation, ongoing erectile aid use, or use of nitrate medications.
* Androgen suppression within the past 6 months or as part of protocol-specified radiotherapy or brachytherapy will be excluded.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Our proposal is aimed at preventing sexual dysfunction and urinary incontinence in prostate cancer survivors, a gender specific cancer.
Enrollment: 12 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahadevan R. Rajasekaran, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Magnetic Stimulation | Sham TPMS
Started | 12 | 0
Completed | 9 | 0
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Prostate cancer survivors with symptoms of urinary incontinence and erectile dysfunction
Groups:
- Magnetic Stimulation: Patients will be subjected to TPMS.
  Sham Magnetic stimulation: Sham Magnetic stimulation for comparison. Despite the pandemic related restrictions during the initial study period, we managed to consent 12 and retain nine patients (age 55-75) for this feasibility study
- Sham TPMS: No patients could be recruited for sham arm
- Total: Total of all reporting groups
Arm/Group | Magnetic Stimulation | Sham TPMS | Total
Number analyzed (Participants) | 12 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants] — Population: Out of the 12 patients consented, only 9 completed the 12-week treatment.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 6 | 0 | 6
    >=65 years | 6 | 0 | 6
Age, Continuous [Mean (Standard Deviation); unit: percentage] — Information is collected using periodic personal interviews and questionnaires.
  percentage | 65 (5) |  | 65 (5)
Sex: Female, Male [Count of Participants; unit: Participants] — The investigators measured symptoms of urine leakage and erectile dysfunction. Population: Out of 12 recruited patients, only 9 completed the 12-week treatment.
  Participants
    Female | 0 | 0 | 0
    Male | 12 | 0 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 6 | 0 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 |  | 12
Patient recruitment [Count of Participants; unit: Participants] | 12 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recruited
Description: Primary outcome measure will be to determine feasibility of recruitment of prostate cancer survivors. We will demonstrate recruitment in VASDHS urology clinics .
Time Frame: During 12-weeks therapy
Population: Prostate cancer survivors with UI and ED.
Measure: Count of Participants; unit: Participants
Groups:
- Magnetic Stimulation: Patients (prostate cancer survivors; with symptoms of urinary incontinence and erectile dysfunction) will be subjected to TPMS.
  Sham Magnetic stimulation: Sham Magnetic stimulation for comparison.
- Sham TPMS: Patients ((prostate cancer survivors; with symptoms of urinary incontinence and erectile dysfunction) will be subjected to sham TPMS
Arm/Group | Magnetic Stimulation | Sham TPMS
Number analyzed (Participants) | 12 | 0
Participants | 12 | 0

2. Primary Outcome: Patient Retention
Description: Retention of these prostate cancer survivors for the study duration.
Time Frame: Retention for 12 week study period.
Population: Prostate cancer survivors with UI and ED.
Measure: Count of Participants; unit: Participants
Arm/Group | Magnetic Stimulation | Sham TPMS
Number analyzed (Participants) | 12 | 0
Participants | 9 |

3. Primary Outcome: Patient Acceptability
Description: Acceptability of TPMS treatment
Time Frame: 12 weeks Post-therapy
Population: Prostate cancer survivors with UI and ED.
Measure: Count of Participants; unit: Participants
Arm/Group | Magnetic Stimulation | Sham TPMS
Number analyzed (Participants) | 9 | 0
Participants | 9 |

4. Secondary Outcome: Number of Participants Who Completed the The International Consultation on Incontinence Questionnaire (ICIQ) to Determine Feasibility to Determine Treatment Outcome
Description: The second objective is to test the feasibility of administering symptom scores in this population to detect severity and early recovery of functional impairment. The investigators will use International Consultation of Incontinence Questionnaire (ICIQ)-symptom score, which assesses the symptoms and effect of UI on quality of life.
Time Frame: 12 weeks post-therapy
Population: Prostate cancer survivors with UI and ED.
Measure: Count of Participants; unit: Participants
Groups:
- Magnetic Stimulation: Patients (prostate cancer survivors; with symptoms of urinary incontinence and erectile dysfunction) will be subjected to TPMS.
  Sham Magnetic stimulation: Sham Magnetic stimulation for comparison. All 12 patients reported that the treatment is acceptable, painless,
- Sham TPMS: Patients (prostate cancer survivors; with symptoms of urinary incontinence and erectile dysfunction) will be subjected to sham TPMS
Arm/Group | Magnetic Stimulation | Sham TPMS
Number analyzed (Participants) | 9 | 0
Participants | 9 | 0

5. Secondary Outcome: Number of Participants Who Completed the The International Index of Erectile Function (IIEF) to Determine Feasibility to Determine Treatment Outcome
Description: The second objective is to test the feasibility of administering symptom scores in this population to detect severity and early recovery of functional impairment. The investigators will evaluate The International Index of Erectile Function (IIEF) symptom scores to test the role of these changes in sexual function symptom severity.
Time Frame: 12 weeks Post-therapy
Population: Prostate cancer survivors with UI and ED.
Measure: Count of Participants; unit: Participants
Arm/Group | Magnetic Stimulation | Sham TPMS
Number analyzed (Participants) | 9 | 0
Participants | 9 |

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the 12-week treatment period.
Description: Patients were asked to report any adverse effect using the Likert scale.
Groups:
- Magnetic Stimulation: Patients (prostate cancer survivors; with symptoms of urinary incontinence and erectile dysfunction) will be subjected to TPMS.
  Sham Magnetic stimulation: Sham Magnetic stimulation for comparison.
  All patients were comfortable with the therapy and reported no adverse effects.
- Sham TPMS: Patients (prostate cancer survivors; with symptoms of urinary incontinence and erectile dysfunction) will be subjected to sham TPMS. No record of any adverse events as there were no patients in this arm.
Arm/Group | Magnetic Stimulation | Sham TPMS
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/0
Other Adverse Events (participants affected / at risk) | 0/12 | 0/0

LIMITATIONS AND CAVEATS:
This is a feasibility study focused on recruitment and retention, and we did not focus on efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT04488068/Prot_SAP_001.pdf
  • Informed Consent Form (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT04488068/ICF_002.pdf